CLINICAL TRIAL: NCT07333313
Title: Study of Oral Uremic Toxin Absorbent/Probiotics to Modulate Systemic Inflammation and Retard the Progression of Chronic Kidney Disease in Patients With Diabetes.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202405001RINE
Record Dates: First submitted 2025-07-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Oral Uremic Toxin Absorbent
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Those who analyze data and those who examine samples are masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral uremic toxin absorbent (Other): Based on these previous findings, we will conduct a prospective randomized open blinded end-point (PROBE) study to see if oral uremic toxin absorbent + probiotics to modulate systemic inflammation and retard the progression of chronic kidney disease in patients with diabetes.
  Interventions: Dietary Supplement: oral uremic toxin absorbent
- probiotics (Other): Based on these previous findings, we will conduct a prospective randomized open blinded end-point (PROBE) study to see if oral uremic toxin absorbent + probiotics to modulate systemic inflammation and retard the progression of chronic kidney disease in patients with diabetes.
  Interventions: Dietary Supplement: probiotics
- oral uremic toxin absorbent +/- probiotics (Experimental): Dietary Supplement: Oral Uremic Toxin Absorbent/Probiotics This 12-month trial will enroll 120 subjects with Diabetic Kidney Disease (DKD), consisting of 60 subjects in CKD Stage 3A, 60 in Stage 3B, 60 in Stage 4, and 60 in Stage 5/dialysis.
  Each group will be randomized into six subgroups (A-F):
  Group A: Administered 2.3g of ABC three times daily during the latter 6 months.
  Group B: Administered 2g of probiotics twice daily during the latter 6 months.
  Group C: Administered a combination of oral uremic toxin absorbent/probiotics during the latter 6 months.
  Clinical evaluations and examinations will be performed at baseline and every 3 months over the 12-month duration, including gut microbiota, inflammatory proteins (e.g., CCL4), long non-coding RNA (lncRNA), and uremic toxins.
  Interventions: Dietary Supplement: oral uremic toxin absorbent + probiotics

INTERVENTIONS:
Dietary Supplement: oral uremic toxin absorbent — In this 12-month trial, 300 DKD participants will be enrolled (60 with CKD stage 3A, 60 with stage 3B, 60 with stage 4, and 60 with stage 5 or on dialysis). Within each stage, participants will be randomized into three subgroups (A-C). Group A will receive ABC 2.3 g three times daily together with standard care during the last 6 months. Group B will receive probiotics 2 g twice daily during the last 6 months. Group C will receive both interventions during the last 6 months. Clinical assessments and examinations- including gut microbiota, inflammatory proteins (e.g., CCL4), long non-coding RNAs (lncRNAs), and uremic toxins- will be conducted at baseline and every 3 months for 12 months.
  Arms: oral uremic toxin absorbent
Dietary Supplement: probiotics — In this 12-month trial, 300 DKD participants will be enrolled (60 with CKD stage 3A, 60 with stage 3B, 60 with stage 4, and 60 with stage 5 or on dialysis). Within each stage, participants will be randomized into three subgroups (A-C). Group A will receive ABC 2.3 g three times daily together with standard care during the last 6 months. Group B will receive probiotics 2 g twice daily during the last 6 months. Group C will receive both interventions during the last 6 months. Clinical assessments and examinations- including gut microbiota, inflammatory proteins (e.g., CCL4), long non-coding RNAs (lncRNAs), and uremic toxins- will be conducted at baseline and every 3 months for 12 months.
  Arms: probiotics
Dietary Supplement: oral uremic toxin absorbent + probiotics — In this 12-month trial, 300 DKD participants will be enrolled (60 with CKD stage 3A, 60 with stage 3B, 60 with stage 4, and 60 with stage 5 or on dialysis). Within each stage, participants will be randomized into three subgroups (A-C). Group A will receive ABC 2.3 g three times daily together with standard care during the last 6 months. Group B will receive probiotics 2 g twice daily during the last 6 months. Group C will receive both interventions during the last 6 months. Clinical assessments and examinations- including gut microbiota, inflammatory proteins (e.g., CCL4), long non-coding RNAs (lncRNAs), and uremic toxins- will be conducted at baseline and every 3 months for 12 months.
  Arms: oral uremic toxin absorbent +/- probiotics

SUMMARY:
Diabetes mellitus (DM) is a chronic inflammatory disease characterized by insufficient insulin secretion or insulin resistance, leading to hyperglycemia. Chronic inflammation and immune system dysfunction are characteristic of DM and can produce a plethora of cytokines and chemokines, thereby contributing to diabetic complications such as cardiovascular events and diabetic vasculopathy in DM. Besides, about 25% of people with diabetes eventually develop diabetic kidney disease (DKD). DKD is a consequence of DM with chronic kidney disease (CKD), which may abruptly increase cardiovascular disease (CVD) and its mortality rate compared with diabetes alone. Therefore, the modulation of the systemic inflammation may have the opportunity to improve both hyperglycemia and diabetic complications including vasculopathy and DKD.

Activated charcoal has been used clinically as a toxin absorbent. Some recent preclinical and clinical observations found the potential benefits and diverse effects of activated charcoal on inflammatory proteins, suggesting its potential immune modulation effects in CKD and related diseases. The current project is then designed to test the hypothesis that oral activated charcoal may be used as an anti-inflammatory strategy for diabetic complications especially DKD. We have recently demonstrated the renal protective effects of a new oral form of non-absorbable activated bamboo charcoal (ABC) in an animal model.

With OMICs studies, a growing preclinical and clinical evidence supports the theory that gut microbiome is a major contributor to adverse cardiovascular outcomes and progression of CKD, and the gut microbiota and its metabolites have the potential to be a novel therapeutic and preventative target for CKD. Additionally, current finding suggests that lncRNAs are involved in cardiovascular (CV) health and diseases. However, there is no report on the impact of gut microbiota on the host circulating lncRNA expression signature and the potential link between gut microbiota, circulating lncRNA levels changes and CKD. Although studies of probiotics which have benefits of CKD patients are numerous, few studies evaluated the effect of coadministration of activated charcoal/probiotics on the patients with CKD.

In this 12-month trial, 120 DKD subjects will be enrolled for each group (CKD group 1: CKD stage 3A; group 2: CKD stage 3B; group 3: CKD stage 4; and group 4: CKD stage 5). Each group of patients will be randomized into 6 subgroups A, B, C, D, E and F. Group A patients will receive ABC 2.3g three times a day in addition to standard care in the first 6 months, but group B patients will receive the same dosage of ABC in the last 6 months. Group C patients will receive probiotics 2g twice a day in addition to standard care in the first 6 months, but group D patients will receive the same dosage of probiotics in the last 6 months. Group E patients will receive ABC 2.3g three times a day and probiotics 2g twice a day in addition to standard care in the first 6 months, but group F patients will receive the same dosage of ABC and probiotics in the last 6 months. All patients will receive clinical assessments and examinations (gut microbiota, inflammatory proteins including CCL4, long-chain noncoding (lnc)RNAs, and uremic toxins) at baseline and every 3 months thereafter for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 years old but not pregnant on the day of screening.
2. DKD patients with stable renal function (Cre elevation < 0.3 mg/dL for at least 30 days) and PCS level (fluctuation < 10% for at least 30 days)
3. Group 1: 120 DKD patients with 45<eGFR<60 ml/min/1.73m2 in stable status. Group 2: 120 DKD patients with 30<eGFR<45 ml/min/1.73m2 in stable status. Group 3: 60 DKD patients with 15<eGFR<30 ml/min/1.73m2 in stable status Group 4: 60 DKD patients with eGFR<15 ml/min/1.73m2 in stable status

Exclusion Criteria:

1. Baseline eGFR > 90 ml/min/1.73m2 according to MDRD equation.
2. Patients in severe malnutrition status, albumin less than 2.0 g/dL.
3. Patients in severe anemia or active gastrointestinal bleeding with hemoglobulin < 8 g/dL.
4. Active peptic ulcer, esophageal varices, ileus or under fasting status
5. Previous gastrointestinal operation.
6. Chronic constipation, as defined with less than 3 bowel movements per week, straining, hard stools.
7. Incomplete evacuation and inability to pass stool. If usage of oral laxatives can achieve bowel movement, this patient will not be excluded.
8. Patients with major hemorrhage, as defined with acute hemorrhage and requirement of blood transfusion during index admission.
9. Patients with a biopsy proved or clinically diagnosed advanced liver cirrhosis, Child classification B or C.
10. Solid organ or hematological transplantation recipients.
11. Evidence of obstructive kidney injury or polycystic kidney disease.
12. Presence or history of malignant neoplasms within the past 5 years prior to the day of screening.
13. Patients with Immune Deficiency Syndrome.
14. Antibiotics or probiotics treatment within the last 3 months before enrollment and during follow-up period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of eGFR | -6th month,-3th month,baseline,random, 3th month and 6th month
  eGFR is estimated GFR calculated by the abbreviated MDRD equation : 186 x (Creatinine/88.4)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if black).

SECONDARY OUTCOMES:
The change of UACR | baseline, 3th month and 6th month
  Urine albumin divided by urine creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital., Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No